CLINICAL TRIAL: NCT02287038
Title: Atomoxetine in Comorbid ADHD/PTSD: A Pilot, Placebo-Controlled Feasibility Study
Brief Title: Atomoxetine in Veterans With Comorbid ADHD/PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1725-P; I01BX007080 (Other Grant/Funding Number: VA Office of Research and Development)
Record Dates: First submitted 2014-10-03; First posted 2014-11-10 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Post Traumatic Stress Disorder; Attention Deficit Hyperactivity Disorder
Keywords: PTSD; ADHD; Atomoxetine; Combat Trauma; Cognitive Deficit
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Attention Deficit Disorder with Hyperactivity; Cognition Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: A small prospective, 10-week, fixed-dose, randomized, double-blind, placebo-controlled, and cross-over trial of atomoxetine as an add-on medication to other therapies in Veterans with comorbid ADHD/PTSD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double-blind, placebo-controlled, and cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atomoxetine 80mg (Active Comparator): Atomoxetine (fixed dose of 80mg), a non-stimulant medication, FDA approve for treatment of ADHD. The active drug will be applied in first phase in group one and in second phase in group two
  Interventions: Drug: Atomoxetine 80 MG
- Placebo (Placebo Comparator): A pharmaceutically inert substance, which will be given to group one in their second phase and group tow in first phase.
  Interventions: Drug: Atomoxetine 80 MG

INTERVENTIONS:
Drug: Atomoxetine 80 MG — Subjects will be randomized and assigned by the study investigator into crossover group 1 (Atomoxetine 80mg at Phase I, then placebo at Phase II) or group 2 (placebo at Phase I, then Atomoxetine at Phase II) with both placebo and medication administered through pharmacy. There was a 1-week interval between the two phases.
  Other Names: Strattera

SUMMARY:
The current available treatments for PTSD are not fully effective for cognitive symptoms of PTSD and have high drop-out and poor engagement, two factors found to be most indicative of overall return to functioning for patients with PTSD. The proposed study directly addresses this knowledge gap by conducting a pilot, fixed-dose, randomized, double-blind, placebo-controlled, and cross-over trial using atomoxetine (ATX) as an add-on medication to other therapies to testing the efficacy of ATX in reducing ADHD cognitive symptoms among veterans with comorbid ADHD/PTSD. Successful completion of this pilot clinical trial may build a platform for future large scale double-blind, placebo-controlled studies using either atomoxetine or other cognitive enhancing medications.

DETAILED DESCRIPTION:
Combat Veterans with posttraumatic stress disorder (PTSD) often show cognitive impairments in attention, working memory, executive functions, and inhibitory control, a cluster of symptoms resembling symptoms of ADHD. The presence of comorbid ADHD cognitive symptoms is often associated with greater PTSD clinical severity and poorer treatment outcomes. While treatments for the avoidance, arousal, and re-experiencing symptoms associated with PTSD for military personnel are readily available, substantial gaps exist in the treatment of the cognitive deficits associated with PTSD. As a result, untreated co-occurring ADHD cognitive symptoms in PTSD may have severe negative impacts on patients' functional recovery, treatment outcome, and quality of life. The proposed study directly addresses this knowledge gap by testing the feasibility and preliminary efficacy of atomoxetine (ATX) in treatment of ADHD cognitive symptoms among those with comorbid ADHD/PTSD. This is a small prospective, 10-week, fixed-dose, randomized, double-blind, placebo-controlled, and cross-over trial of ATX as an add-on medication to other therapies in Veterans with comorbid ADHD/PTSD. Primary outcome measures will be ADHD cognitive symptom reduction and quality of life improvement as measured by the Adult ADHD Rating Scales-Self-Report: Short Version (CAARS-S:S) and the Adult ADHD Quality of Life-29 (AAQoL-29). Secondary outcome measures will be PTSD and depressive symptoms reduction as measured by the Clinician Administered PTSD Scale (CAPS), the Hamilton Depression Scale (HAM-D). In addition to subjective measures, the response inhibition task Go/NoGo (GNG) will be used as objective assessments to measure ATX treatment outcomes. The proposed work is innovative; it applies novel therapeutic agent to treat cognitive symptoms in PTSD. To our knowledge, this is the first study to apply a SNRI to address an often overlooked PTSD-cognitive deficit. This study is directly responsive to the mission of RR&D-SPiRE "to maximize functional recovery" of cognitive function in PTSD. The outcome of the proposed research will be significant, because it provides a knowledge base to help determine who is at risk for developing treatment resistance among PTSD patients, thereby allowing for development of early intervention strategies. More importantly, this clinical trial may immediate benefit Veterans by enhancing their cognitive function, reducing ADHD symptoms related disability, and further improving quality of life for veterans suffer from comorbid ADHD/PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 20 to 60 with PTSD and significant ADHD symptoms (CAARS-S:S > 65);
* Good physical health.
* Evidence of combat as defined by:

  * Trauma exposure sufficient to meet Category A of PTSD criteria (Breslau and Kessler 2001)

Exclusion Criteria:

* Age younger than 20 or greater than 60.
* Known sensitivity to ATX
* Presence of disorders that could conceivable be exacerbated by atomoxetine (specifically, narrow angle closure glaucoma, urinary outflow obstruction, hypertension, and neurological disorders, particularly tics and Tourette's syndrome, or a history of epilepsy or seizures).
* Use of concomitant medication that could potentially interact with atomoxetine including monoamine oxidase inhibitors (MAOI), antihypertensive medication, or any concomitant medication that was a cytochrome 2D6 inhibitor (CYP2D6), since atomoxetine's elimination involves the CYP2D6 system.
* An active or lifetime major mental health diagnosis as determined by DSM-IV Axis I Disorders, including schizophrenia, schizoaffective disorder, psychotic disorder not otherwise specified, bipolar I disorder, bipolar II disorder, bipolar disorder not otherwise specified. The project will allow presence of depressive disorders if the depressive episodes are secondary to PTSD.
* Current substance dependence and abuse (within 3 month).
* Females who are pregnant.
* Suicidal thoughts and behavior. b. Sources of Material

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhewu Wang, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Zuschlag ZD, Myers US, Hamner M. Atomoxetine in comorbid ADHD/PTSD: A randomized, placebo controlled, pilot, and feasibility study. Depress Anxiety. 2022 Apr;39(4):286-295. doi: 10.1002/da.23248. Epub 2022 Mar 21. PMID 35312136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants are explained the nature, purpose, and procedure of the study and asked to sign an informed consent that will explain the potential risks and benefits of the study participation. Primary, secondary outcome measures, and physical examination will be conducted at baseline and all subsequent visits by a qualified research clinician.
Pre-assignment Details: Week 1: Screening; Week 2 to 5: Phase 1 (ATX in group 1 and placebo in group2); Week 6: Wash-out; Week 7 to 10: Phase 2 (Crossover, Placebo in group1 and ATX in group2).
Groups:
- Group 1. Atomoxitine First, Then Placebo: Subjects in Group 1: First Intervention (4 weeks with Atomoxetine), Wash-out (1 week), and Second Intervention (4 weeks with placebo)
- Group 2. Placebo First, Then Atomoxitine: Subjects in Group 1: First Intervention (4 weeks with placebo), Wash-out (1 week), and Second Intervention (4 weeks with Atomoxetine)
Period: Overall Study
Arm/Group | Group 1. Atomoxitine First, Then Placebo | Group 2. Placebo First, Then Atomoxitine
Started | 23 | 21
Completed | 18 | 18
Not Completed | 5 | 3
Not completed — Stopped attending appointments | 3 | 2
Not completed — Anxiety after starting medication | 0 | 1
Not completed — Nausea after starting medication | 1 | 0
Not completed — Abnormal ECG after starting medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group1: Group 1: Atomoxetine during the first phase ( 4 Weeks), the Wash-out (1week), followed by a second phase (4 Weeks) of placebo.
- Group 2: Group 2: Placebo during the first phase ( 4 Weeks), the Wash-out (1week), followed by a second phase (4 Weeks) of Atomoxetine.
- Total: Total of all reporting groups
Arm/Group | Group1 | Group 2 | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Customized [Mean (Full Range); unit: years] | 41.2 [30 to 53] | 41.0 [24 to 59] | 41 [24 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 23 | 20 | 43
  Unknown or Not Reported | 0 | 0 | 0
CAARS-S:S [Mean (Standard Deviation); unit: units on a scale] — The CAARS-S:S is a 26-item questionnaire that assesses symptoms of ADHD in persons aged 18 years or older. T-scores above 65 indicate a likelihood of moderate to severe ADHD symptoms and impairment. The range for the CAARS-S:S is from 0 to 78. A score of 78 would resemble the worst symptoms of ADHD with a score 0 having no symptoms. This measurement can be used for both diagnostic and symptoms severity evaluations. Therefore it is used both in screening and follow up visits. Population: The study analyzed 36 participants. 8 participants dropped out of the study.
  units on a scale
    number analyzed (Participants) | 18 | 18 | 36
    (all) | 74.78 (9.54) | 69.33 (9.89) | 72.06 (9.97)

OUTCOME MEASURES:

1. Primary Outcome: Conners' Adult ADHD Rating Scales-Self-Report: Short Version (CAARS-S:S, Conner et al, 1999)
Description: Conners' Adult ADHD Rating Scales-Self-Report: Short Version (CAARS-S:S, Conner et al, 1999): The CAARS-S:S is a 26-item questionnaire that assesses symptoms of ADHD in persons aged 18 years or older. T-scores above 65 indicate a likelihood of moderate to severe ADHD symptoms and impairment. The range for the CAARS-S:S is from 0 to 78. A score of 78 would resemble the worst symptoms of ADHD with a score 0 having no symptoms.
Time Frame: Visit 1, (Day1), Visit 4(Day 36), Visit 7 (Day 71)
Population: The 36 patients that completed at least one phase of the study were included in the final analyses. The 8 participants did not finish the first phase, and data were not collected on those 8 subjects on the week 4 and week 7. Therefore, the 8 subjects were not entered to the final analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm1: Atomoxetine: This is a crossover study in which the participants would receive Atomoxetine and Placebo. Group 1 received Atomoxetine during the first phase, and Group2 receive Atomoxetine in the second phase.
- Arm 2: Placebo: This is a crossover study in which the participants would receive Atomoxetine and Placebo. Group 2 received the placebo during the first phase, and Group 1 receive placebo during the second phase.
Arm/Group | Arm1: Atomoxetine | Arm 2: Placebo
Number analyzed (Participants) | 36 | 36
units on a scale
  Before the intervention | 75.12 (9.23) | 68.56 (9.34)
  After the intervention | 67.79 (8.79) | 72.80 (8.91)

2. Primary Outcome: The Adult ADHD Quality of Life-29 (AAQOL-29, Brod et al, 2006)
Description: The Adult ADHD Quality of Life-29 (AAQOL-29, Brod et al, 2006): AAQoL-29 is a 29-item questionnaire designed to assess quality of life and was a secondary efficacy measure in this trial. It is a participant-reported outcome measure used to examine disease specific functional impairments and quality of life for adults with ADHD. The AAQoL is scored as an overall total score, measuring Life Productivity, Psycholofical Health, Relationship, and Life Outlook. Each item is rated by patients on a 5-point Likert scale ranging from "Not at all/Never" (1) to "Extremely/Very Often" (5). To derive overall scores, item scores are transformed to a 0-100-point scale (1=0; 2=25; 3=50; 4=75; 5=100). Then, the item scores are summed up and divided by item count to generate overall scores. The score range from 0 to 100. A higher score indicates greater QoL and better functioning.
Time Frame: Visit 1 (Day1), 4(Day 36), 7 (Day 71)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Atomoxetine: This is a crossover study in which the participants would receive Atomoxetine and Placebo. Group 1 will receive Atomoxetine during the first phase and Group 2 would receive Atomoxetine in the second phase.
- Arm 2: Placebo: This is a crossover study in which the participants would receive Atomoxetine and Placebo. Group 2 will receive placebo during the first phase and Group 1 would receive placebo in the second phase.
Arm/Group | Arm 1: Atomoxetine | Arm 2: Placebo
Number analyzed (Participants) | 36 | 36
units on a scale
  Before intervention | 33.61 (11.52) | 36.51 (11.18)
  After Intervention | 43.51 (9.80) | 37.23 (11.12)

ADVERSE EVENTS:
Time Frame: The adverse events were monitored at Week 2 (Day14, Visit 2), week 5 (Day 36, Visit 4), and week 9 (Day 71, Visit 7).
Description: Nausea and Anxiety after starting medication were reported by some of the participants, Majority of participants who had minor Nausea were able to finish the trial. However, two participants dropped out due to Nausea and Anxiety. The two drop out participants were followed up and no further adverse reaction were observed after discontinuation of the trial. One participant had EKG abnormality at screen, and the participant withdraw before the trial.
Groups:
- Arm1, Atomoxetine: Group 1 received Atomoxetine during the first phase of the study, and Group 2 received Atomoxetine during the second phase.
- Arm2, Placebo: Group 2 received the placebo during the first phase of the study, and Group 1 received the placebo during the second phase.
Arm/Group | Arm1, Atomoxetine | Arm2, Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 2/36 | 0/36
OTHER ADVERSE EVENTS (reported when occurring in more than 2.28% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm1, Atomoxetine (N=36) | Arm2, Placebo (N=36)
Nausea after starting medication (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anxiety after starting medication (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02287038/Prot_SAP_000.pdf